CLINICAL TRIAL: NCT04880720
Title: Deciphering a Specific Signature of the Immunosenescence Induced in COVID-19+ Patients Versus Rheumatoid Arthritis Patients
Acronym: SENO-COVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0454
Record Dates: First submitted 2021-05-10; First posted 2021-05-11 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: SARS-Cov-2 Infection; Rheumatoid Arthritis
MeSH Terms: conditions — COVID-19; Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 Patients
  Interventions: Other: Blood sampling
- Rheumatoid Arthritis Patients
  Interventions: Other: Blood sampling
- Healthy Comparator
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling - 10mL

SUMMARY:
Immune aging or immunosenescence is characterized by a loss of T cell clonal diversity and a contraction of naïve T cells with proliferative capacity associated with the functional impairment of many others immune cells as well as a chronic low degree of inflammation. A restrictive T cell repertoire is likely more prone to antigen-mediated exhaustion observed during chronic viral infections. Notably, lymphopenia is the most consistent laboratory abnormality in COVID-19 infected patients and both lung-resident and circulating T cells potently up-regulate markers of T cell exhaustion. It is not clear today if the association of COVID-19 disease severity with age is mainly related with the immunosenescence of infected patients. Interestingly, T cell exhaustion and premature immunosenescence have also been observed in chronic inflammatory diseases such as rheumatoid arthritis (RA). To better understand the immunological mechanisms involved in SARS-Cov-2 pathophysiology, the investigators propose to compare the immunosenescence patterns observed during RA, aging and SARS-Cov-2 infected patients in order to design improved therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria for Active RA Patients:

* Patients with rheumatoid arthritis (RA) meeting the 2010 ACR/EULAR diagnostic criteria
* Patients in inflammatory flare of RA (DAS28 > 3.2)
* Patients who have been off biological disease-modifying antirheumatic drugs (bDMARDs) or targeted synthetic antirheumatic drugs (tsDMARDs) for RA for at least 2 weeks (except for rituximab, where a delay of at least 12 months is required)
* Conventional synthetic DMARDs (Methotrexate, Hydroxychloroquine, Leflunomide, Sulfasalazine) are allowed
* Beneficiary of a social security system
* Informed consent

Inclusion Criteria for Healthy Controls:

* Absence of chronic diseases and current infection
* Beneficiary of a social security system
* Informed consent

Inclusion Criteria for COVID-19+ Patients:

* Patients with ongoing SARS-Cov-2 infection (PCR+)
* Patients hospitalized at D7-D14 of symptoms onset
* Patients with two or more SARS-Cov-2 symptoms (including fever, cough, dyspnea, sore throat, chest pain, anosmia, diarrhea)
* Membership in or beneficiary of a social security scheme
* Collection of free and informed consent

Exclusion Criteria for All Groups:

* Subjects under 18 years of age
* HIV positive patients
* Diabetic patients
* Morbidly obese patients (BMI > 40kg/m2)
* Use of senolytic drugs in the week prior to inclusion (azithromycin, metformin, cyclosporine, JAK inhibitors)
* Use of steroids in doses greater than 10 mg/day in the week prior to inclusion
* Subjects unable to give consent
* Pregnant, breastfeeding, or non-menopausal women not taking effective contraception
* Vulnerable subjects protected by law
* Subjects under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * COVID-19 patients are recruited through the Covidothèque project and the UANDES center (Chile)
  * RA patients and healthy subjects are recruited through 3 rheumatology reference centers (Montpellier, Paris Saint-Antoine and Saint-Etienne)
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Results of phenotypic immunosenescence analyses of COVID-19 patients targeting 5 different immune populations (neutrophils, T lymphocytes, NK lymphocytes, B lymphocytes and monocytes). | At inclusion visit

SECONDARY OUTCOMES:
Comparison of previous results with the results of senescence immunophenotyping in peripheral blood of a reference population with an inflammatory disease (active RA) | At inclusion visit
Comparison of previous results with the results of senescence immunophenotyping in peripheral blood of a reference population of healthy controls. | At inclusion visit
Identification of a specific gene expression of immunosenescence induced in COVID-19 patients, using transcriptomic analysis in the different immune subpopulations previously identified and specific to COVID-19 patients. | At inclusion visit

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

REFERENCES:
- [Background] Wang R, Pan M, Zhang X, Han M, Fan X, Zhao F, Miao M, Xu J, Guan M, Deng X, Chen X, Shen L. Epidemiological and clinical features of 125 Hospitalized Patients with COVID-19 in Fuyang, Anhui, China. Int J Infect Dis. 2020 Jun;95:421-428. doi: 10.1016/j.ijid.2020.03.070. Epub 2020 Apr 11. PMID 32289565
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Li X, Xu S, Yu M, Wang K, Tao Y, Zhou Y, Shi J, Zhou M, Wu B, Yang Z, Zhang C, Yue J, Zhang Z, Renz H, Liu X, Xie J, Xie M, Zhao J. Risk factors for severity and mortality in adult COVID-19 inpatients in Wuhan. J Allergy Clin Immunol. 2020 Jul;146(1):110-118. doi: 10.1016/j.jaci.2020.04.006. Epub 2020 Apr 12. PMID 32294485
- [Background] Rockx B, Baas T, Zornetzer GA, Haagmans B, Sheahan T, Frieman M, Dyer MD, Teal TH, Proll S, van den Brand J, Baric R, Katze MG. Early upregulation of acute respiratory distress syndrome-associated cytokines promotes lethal disease in an aged-mouse model of severe acute respiratory syndrome coronavirus infection. J Virol. 2009 Jul;83(14):7062-74. doi: 10.1128/JVI.00127-09. Epub 2009 May 6. PMID 19420084
- [Background] Maringer K, Fernandez-Sesma A. Message in a bottle: lessons learned from antagonism of STING signalling during RNA virus infection. Cytokine Growth Factor Rev. 2014 Dec;25(6):669-79. doi: 10.1016/j.cytogfr.2014.08.004. Epub 2014 Aug 24. PMID 25212897
- [Background] Nikolich-Zugich J. The twilight of immunity: emerging concepts in aging of the immune system. Nat Immunol. 2018 Jan;19(1):10-19. doi: 10.1038/s41590-017-0006-x. Epub 2017 Dec 14. PMID 29242543
- [Background] Fulop T, Larbi A, Dupuis G, Le Page A, Frost EH, Cohen AA, Witkowski JM, Franceschi C. Immunosenescence and Inflamm-Aging As Two Sides of the Same Coin: Friends or Foes? Front Immunol. 2018 Jan 10;8:1960. doi: 10.3389/fimmu.2017.01960. eCollection 2017. PMID 29375577
- [Background] Tachikart Y, Malaise O, Mumme M, Jorgensen C, Brondello JM. Seno-suppressive molecules as new therapeutic perspectives in rheumatic diseases. Biochem Pharmacol. 2019 Jul;165:126-133. doi: 10.1016/j.bcp.2019.03.017. Epub 2019 Mar 13. PMID 30878551
- [Background] Oh SJ, Lee JK, Shin OS. Aging and the Immune System: the Impact of Immunosenescence on Viral Infection, Immunity and Vaccine Immunogenicity. Immune Netw. 2019 Nov 14;19(6):e37. doi: 10.4110/in.2019.19.e37. eCollection 2019 Dec. PMID 31921467
- [Background] Vicente R, Mausset-Bonnefont AL, Jorgensen C, Louis-Plence P, Brondello JM. Cellular senescence impact on immune cell fate and function. Aging Cell. 2016 Jun;15(3):400-6. doi: 10.1111/acel.12455. Epub 2016 Feb 22. PMID 26910559
- [Background] Campos C, Pera A, Sanchez-Correa B, Alonso C, Lopez-Fernandez I, Morgado S, Tarazona R, Solana R. Effect of age and CMV on NK cell subpopulations. Exp Gerontol. 2014 Jun;54:130-7. doi: 10.1016/j.exger.2014.01.008. Epub 2014 Jan 17. PMID 24440462
- [Background] Appay V, Almeida JR, Sauce D, Autran B, Papagno L. Accelerated immune senescence and HIV-1 infection. Exp Gerontol. 2007 May;42(5):432-7. doi: 10.1016/j.exger.2006.12.003. Epub 2007 Jan 8. PMID 17307327
- [Background] Goronzy JJ, Lee WW, Weyand CM. Aging and T-cell diversity. Exp Gerontol. 2007 May;42(5):400-6. doi: 10.1016/j.exger.2006.11.016. Epub 2007 Jan 10. PMID 17218073
- [Background] Lin L, Lu L, Cao W, Li T. Hypothesis for potential pathogenesis of SARS-CoV-2 infection-a review of immune changes in patients with viral pneumonia. Emerg Microbes Infect. 2020 Dec;9(1):727-732. doi: 10.1080/22221751.2020.1746199. PMID 32196410
- [Background] de Wit E, van Doremalen N, Falzarano D, Munster VJ. SARS and MERS: recent insights into emerging coronaviruses. Nat Rev Microbiol. 2016 Aug;14(8):523-34. doi: 10.1038/nrmicro.2016.81. Epub 2016 Jun 27. PMID 27344959
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] D'Antiga L. Coronaviruses and Immunosuppressed Patients: The Facts During the Third Epidemic. Liver Transpl. 2020 Jun;26(6):832-834. doi: 10.1002/lt.25756. Epub 2020 Apr 24. No abstract available. PMID 32196933
- [Background] Giacalone VD, Margaroli C, Mall MA, Tirouvanziam R. Neutrophil Adaptations upon Recruitment to the Lung: New Concepts and Implications for Homeostasis and Disease. Int J Mol Sci. 2020 Jan 28;21(3):851. doi: 10.3390/ijms21030851. PMID 32013006
- [Background] Biswas SK, Mantovani A. Macrophage plasticity and interaction with lymphocyte subsets: cancer as a paradigm. Nat Immunol. 2010 Oct;11(10):889-96. doi: 10.1038/ni.1937. Epub 2010 Sep 20. PMID 20856220
- [Background] Nicolas-Avila JA, Adrover JM, Hidalgo A. Neutrophils in Homeostasis, Immunity, and Cancer. Immunity. 2017 Jan 17;46(1):15-28. doi: 10.1016/j.immuni.2016.12.012. PMID 28099862
- [Background] Cloke T, Munder M, Bergin P, Herath S, Modolell M, Taylor G, Muller I, Kropf P. Phenotypic alteration of neutrophils in the blood of HIV seropositive patients. PLoS One. 2013 Sep 9;8(9):e72034. doi: 10.1371/journal.pone.0072034. eCollection 2013. PMID 24039734
- [Background] Bowers NL, Helton ES, Huijbregts RP, Goepfert PA, Heath SL, Hel Z. Immune suppression by neutrophils in HIV-1 infection: role of PD-L1/PD-1 pathway. PLoS Pathog. 2014 Mar 13;10(3):e1003993. doi: 10.1371/journal.ppat.1003993. eCollection 2014 Mar. PMID 24626392
- [Background] Li X, Geng M, Peng Y, Meng L, Lu S. Molecular immune pathogenesis and diagnosis of COVID-19. J Pharm Anal. 2020 Apr;10(2):102-108. doi: 10.1016/j.jpha.2020.03.001. Epub 2020 Mar 5. PMID 32282863
- [Background] Qin C, Zhou L, Hu Z, Zhang S, Yang S, Tao Y, Xie C, Ma K, Shang K, Wang W, Tian DS. Dysregulation of Immune Response in Patients With Coronavirus 2019 (COVID-19) in Wuhan, China. Clin Infect Dis. 2020 Jul 28;71(15):762-768. doi: 10.1093/cid/ciaa248. PMID 32161940
- [Background] Zheng M, Gao Y, Wang G, Song G, Liu S, Sun D, Xu Y, Tian Z. Functional exhaustion of antiviral lymphocytes in COVID-19 patients. Cell Mol Immunol. 2020 May;17(5):533-535. doi: 10.1038/s41423-020-0402-2. Epub 2020 Mar 19. No abstract available. PMID 32203188